CLINICAL TRIAL: NCT02347501
Title: Dipeptidyl Peptidase-4 Inhibition and Narrow-band Ultraviolet-B Light in Psoriasis (DINUP): A Randomised Clinical Trial
Brief Title: Dipeptidyl Peptidase-4 Inhibition and Narrow-band Ultraviolet-B Light in Psoriasis (DINUP)
Acronym: DINUP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPIP-2012-02; 2012-005483-10 (EudraCT Number)
Record Dates: First submitted 2015-01-13; First posted 2015-01-27 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Sitagliptin 100mg once daily orally or 50mg once daily for participants with moderate kidney disease for 24 weeks and narrowband ultraviolet-B (NBUVB) phototherapy.
  NBUVB light therapy is continued until the participants' psoriasis clears (<1% body surface area involved).
  Interventions: Drug: Sitagliptin (Januvia)
- B (No Intervention): No additional treatment other than narrowband ultraviolet-B (NBUVB) phototherapy.
  NBUVB light therapy is continued until the participants' psoriasis clears (<1% body surface area involved).

INTERVENTIONS:
Drug: Sitagliptin (Januvia) — Sitagliptin 100mg tablet once daily (or 50mg once daily for participants with moderate kidney disease) for twenty four weeks in patients due to undergo NBUVB light therapy.
  Other Names: Januvia
  Arms: A

SUMMARY:
The primary purpose of this study is to determine if sitagliptin (Januvia®) improves psoriasis severity after 24 weeks of treatment in 60 participants with psoriasis who do not have type 2 diabetes mellitus, and who are due to receive a course of narrowband ultraviolet-B phototherapy (NB-UVB). The investigators will compare the change in psoriasis severity in 60 participants treated with both sitagliptin and NB-UVB to 60 participants treated with NB-UVB alone. Participants will be recruited from two centres and after a 3 week run-in period will be followed prospectively for 36 weeks. Participants will be stratified by centre, plasma glycated haemoglobin level (HbA1c), obesity status and previous response to NB-UVB, after which they will be randomly allocated to Arm A or Arm B. Participants will be treated with either sitagliptin for 24 weeks and NB-UVB (Arm A), or NB-UVB alone (Arm B).

Both the research participants and the investigators will be aware of the trial arm to which the research participant has been allocated randomly (open-label study). Research participants are prohibited from using systemic psoriasis therapy for the duration of their trial involvement.

Participants will be assessed at 8 study visits over 39 weeks. Participants will complete questionnaires, have a medical history recorded and physical examination, blood sampling and skin biopsies taken (in a small number of willing participants at 2 visits).

The following endpoints will be analysed:

Changes in psoriasis severity at 24 and 36 weeks; changes in validated quality of life scores; incidence of adverse events; incidence of discontinuation of one of the study IMPs, time to relapse of psoriasis; changes in cardiovascular disease risk factor profiles; changes in cytokines, hormones, expression of immune proteins in blood and skin biopsies; and genetic profiles that predicts best response to sitagliptin therapy.

The investigators hypothesize that sitagliptin therapy decreases psoriasis severity.

DETAILED DESCRIPTION:
Background:

Psoriasis is a chronic, autoimmune skin disease affecting approximately 2% of the world's population. It is characterised by keratinocyte hyperproliferation, by aberrant keratinocyte differentiation and by cutaneous inflammation.

Dipeptidyl peptidase-4 (DPP-4) is expressed on keratinocytes and its activity is upregulated in psoriasis. DPP-4 inhibition suppresses keratinocyte proliferation and restores partially keratinocyte differentiation. The main site of DPP-4 activity is cluster of differentiation antigen 26 (CD26). CD26 is a marker of T cell activation and is a key molecule in the pathogenesis of autoimmune diseases. One case of DPP-4 inhibitor therapy improving psoriasis severity has been reported.

Agents used to treat psoriasis target commonly the underlying inflammation. C-reactive protein (CRP) is a sensitive, systemic marker of inflammation. In people with type 2 diabetes (T2DM) DPP-4 inhibitor therapy decreases CRP concentrations. Serum CRP concentrations correlate with psoriasis severity and interventions that decrease the CRP concentration may decrease also psoriasis severity. Medications that improve insulin resistance may decrease also systemic inflammation and improve psoriasis. We have shown previously, in psoriasis patients without T2DM (both lean and obese), that the fasting insulin concentration and the homeostatic model of insulin resistance (measures of insulin resistance) correlate strongly with the psoriasis area and severity index (PASI, a measure of psoriasis severity: r=0.48, p<0.001; r=0.49, p<0.001).

DPP-4 inhibitors prevent also the degradation of insulin secretagogues, such as glucagon-like peptide-1 (GLP-1), thereby ameliorating hyperglycaemia without causing hypoglycaemia. Due to this effect DPP-4 inhibitors are effective for the treatment of T2DM. Other interventions which increase GLP-1 receptor activation, such as roux-en-Y gastric bypass surgery and GLP-1 analogue therapy, can improve also psoriasis severity.

We have reported previously a significant improvement in two patients with psoriasis and diabetes treated with the GLP-1 analogue liraglutide. In a subsequent open study of 7 patients with both psoriasis and type 2 diabetes we found a significant reduction in psoriasis severity and a significant improvement in quality of life following treatment with liraglutide.

Name and Description of the Investigational Medicinal Products(s):

Januvia® 100 mg tablets, which are film-coated tablets for oral ingestion that contain 100mg of the dipeptidyl peptidase-4 inhibitor sitagliptin.

For research participants with moderate kidney disease (CrCl < 50 ml/min or eGFR < 50 ml/min/1.73m2), a dose of 50mg per day of sitagliptin will be used.

Potential risks and benefits:

More than 1% of people who take Januvia® tablets experience upper respiratory tract infection (no greater incidence than with placebo), hypoglycaemia (no greater incidence than with placebo), headache or limb pain.

The potential benefits of DPP-4 inhibition include decreased risk of cardiovascular disease and decreased risk of bone fracture.

The anticipated benefits of Januvia® therapy in psoriasis patients without type 2 diabetes thus justify the potential risks.

Description of and justification for the route of administration, dosage, dosage regimen and treatment period:

This will be a two centre, thirty-nine week, prospective, randomized, open-label clinical trial of oral Januvia® (sitagliptin) tablets in 120 people with psoriasis without diabetes who are due to undergo a course of NB-UVB phototherapy.

After a three week run-in period, where research participants will not receive the investigational medicinal product, research participants will be allocated randomly, after stratification by centre, by HbA1c level (HbA1c < 38mmol/mol or ≥ 38mmol/mol), BMI level (BMI < 30 kg/m2 or ≥ 30 kg/m2) and previous response to NB-UVB (achieved remission within 25 exposures during most recent course of NBUVB or not) either to Arm A or to Arm B. Those who have not been exposed previously to NBUVB will be placed in the "did not achieve remission within 25 exposures" group. Research participants allocated to Arm A will receive a twenty six week supply of Januvia® tablets (DPP-4 Inhibitor) and will be instructed to ingest orally one 100mg tablet once daily (or 50mg once daily for participants with moderate kidney disease) for twenty four weeks. Research participants allocated to Arm B will receive no treatment (aside from usual medications and phototherapy). Both the research participants and the investigators will be aware of the trial arm to which the research participant has been allocated randomly (open-label study).

Research participants will be prohibited from making any changes to the dose of medications used to treat psoriasis. Any other medications that are considered necessary for the participant's welfare and will not interfere with the study medication may be given at the discretion of the Investigator.

Januvia® is licensed to improve glycaemic control for people with type 2 diabetes (T2DM). The Summary of Product Characteristics (SPC) states that the dose of Januvia® is 100mg once daily (using tablets for oral ingestion). For research participants with moderate kidney disease (CrCl < 50 ml/min or eGFR < 50 ml/min/1.73m2), the Summary of Product Characteristics (SPC) states that the dose of Januvia® is 50mg once daily (using tablets for oral ingestion). In keeping with this all participants with an eGFR < 50ml/min/1.73m2 who are due to receive Januvia® will receive 50mg once daily.

Study Hypothesis:

Dipeptidyl peptidase-4 inhibitor therapy decreases psoriasis severity.

Statement of Trial Conduct:

This trial will be conducted in compliance with the protocol, with the guidelines of the Declaration of Helsinki (see Appendix 2), with the International Conference of Harmonisation Tripartite Guideline on Good Clinical Practice, with all applicable regulatory requirements and with data protection legislation (Data Protection Act 1988 and Data Protection Amendment Act 2003)

Cohort:

The population to be studied will be psoriasis patients with type 2 diabetes.

We plan to enrol 120 research participants in total. Research participants will be recruited from two centres: St Vincent's University Hospital, Elm Park, Dublin 4 and Adelaide and Meath Hospital, Tallaght, Dublin 24. These hospitals provide outpatient dermatology services. Psoriasis patients attending these centres who have a psoriasis area and severity index (PASI) greater than 7 and who are due to undergo a course of NB-UVB phototherapy will be considered potentially eligible research participants and will be invited to attend for a screening visit.

Identification and Recruitment:

Potentially eligible research participants will be identified through use of patient databases in St Vincent's University Hospital and in Adelaide and Meath Hospital and through review of healthcare records in St Vincent's University Hospital and in Adelaide and Meath Hospital.

Potentially eligible research participants will be recruited in one of two ways by the study investigators or suitably qualified designee. One of these two ways will be during a clinic visit by the study investigators or suitably qualified designee. The other of the two ways will be mailing a letter of invitation.

A record of all medication taken by study participants in the month before visit 1 and concomitant medication a participant takes throughout the study will be recorded on the appropriate page of the Case Report Form (CRF).

Treatment compliance of research participants will be measured by pill counts. Research participants will be instructed to bring opened, unopened and empty investigational medicinal product packages to each visit in order to allow the assessment of compliance with study treatment. A record of all investigational medicinal product dispensed and returned will be documented on the investigational medicinal product dispensing and accountability log. Blood taken during stages when the participant is expected to be taking drug therapy will be used for future determination of plasma glucose and glycated haemoglobin concentrations. These concentrations will also be used to help ascertain compliance with the allocated treatment regimen.

Blood samples for measurement of laboratory parameters will be taken between the hours of 0800 and 1200 after a greater than 12 hour overnight fast (with the exception of the Screening Visit when participants can attend in a non fasting state) and before ingestion of the study investigational medicinal product. The blood will be taken by a senior clinician, or suitably qualified designee, with competence and experience in the procedure of venepuncture.

Thirty millilitres (30ml) of blood will be drawn during visit 1, and 73.5 ml during visit 2. Sixty millilitres (60ml) of blood will be drawn from the research participants during visits 3 to 5, and at visit 7. During visits 6 and 8, 67.5 mls of blood will be drawn.Blood will be drawn into vacutainer tubes containing either ethylenediaminetetraacetic acid (EDTA), lithium heparin, sodium fluoride, clot activator or a DPP-4 inhibitor cocktail.

Each research participant will be asked to give a blood sample for genetic analysis at the 2nd Visit. These genetic samples will be analysed to try determine the genetic, and/or epigenetic, profile that predicts best response to DPP-4 inhibitor therapy.

Whole blood will be stored for future DNA extraction using the protocols detailed in the Molecular Medicine Ireland Guideline for Standardised Biobanking (First Edition 2010). This involves drawing blood into a blood tube containing EDTA and storing the blood tube at -20°C in secure, dedicated freezers in the Research Laboratories in the Education and Research Centre in St Vincent's University Hospital. The blood will be stored within 12 hours of blood collection.

Blood that has been stored for future DNA extraction will be destroyed once the DNA analyses are complete. Disposal of this material will be in accordance with current practice in this unit and with the written protocols in place in this unit. Disposal will involve the use of solid plastic waste containers which will be sent for incineration.

To protect the research participant's identity, a unique identification code will be assigned by the Investigator, or authorised designee, to each participant's genetic sample and used in lieu of the participant's name. This coded form of identification, instead of the participant's name, will appear on all documents/databases.

Statistical Analysis Plan:

Demographic and baseline clinical data will be summarized using descriptive statistics by treatment group. Similarly, the primary and secondary efficacy variables will be summarized using descriptive statistics by treatment group.

Data from research participants who are not allocated to either arm of the study and who do not receive a supply of the investigational medicinal product will be excluded from statistical analyses.

T tests (or the appropriate alternative for non-parametric data), using two-sided tests, will be used to test for significant differences between the sets of data obtained. The independent samples T test will be used to assess for differences between the effects of the test product (Januvia®) compared to the effects of no additional treatment. Chi square analyses will be used to test for significant differences in categorical variables between the sets of data obtained.

Subgroup analyses will be performed on those research participants who:

complete the visit 6 assessment; have severe psoriasis; have non-severe psoriasis; are male; are female; are obese; and are older than 45 years.

Packaging and Labelling:

All study medication will be labelled and stored in accordance with Annex 13 of the EU guidelines of good manufacturing practice in respect of investigational medicinal products for human use, the SPC and hospital procedures.

Screening visit (Visit 1, Week -3) Before any screening examinations take place potentially eligible research participants will be given a full explanation as to what participation in the study would involve - this will be done both verbally and in writing in the form of a written participant information leaflet. Potential research participants will be given sufficient time to consider their participation in the study and to ask any questions concerning the study. Potential research participants who are willing to take part in the study will be asked then to sign an informed consent form. No study related procedures will take place for any research participant before the informed consent form has been signed.

The following assessments will then be performed:

1. Checking against inclusion and exclusion criteria;
2. Obtaining demographic information;
3. Obtaining a detailed medical history (previously diagnosed illnesses etc);
4. Obtaining a detailed medication history for the previous month;
5. Measurement of weight, blood pressure and heart rate;
6. Performing a urine based pregnancy test (women of child bearing potential only);
7. Assessment of PASI; and
8. Blood sampling for laboratory examination.

An identification number will be allocated to the potential research participant following informed consent and provided that he or she meets the inclusion criteria and does not have an exclusion criterion to study entry. This identification number, together with the participant's initials, will act as a unique identifier for that participant.

Baseline (Visit 2, Day 0) The potential research participant will return for the baseline visit within three weeks of the screening visit.

The following assessments will be performed:

1. Completion of quality of life questionnaires by the research participant (Dermatology Life Quality Index (DLQI); EuroQol five item questionnaire (EQ-5D); Hospital Anxiety and Depression Scale (HADS); and Stanford HAQ 8-Item Disability Scale (HAQ-8) ;
2. Recording of adverse events;
3. Recording of changes in concomitant medication;
4. Measurement of height, weight, blood pressure and heart rate;
5. Performing a urine based pregnancy test (women of child bearing potential only);
6. Assessment of PASI; and
7. Blood sampling for laboratory examination. If the participant is willing a skin biopsy will be performed, using a sterile technique by an experienced physician, to determine skin immune cell number and skin pro-inflammatory protein level.

If a participant is noted to score greater than 8 (out of 21) on either the anxiety or the depression components of the HADS, at this or any subsequent study visits, their General Practitioner (GP) will be advised of this and of the high likelihood of depressive/affective mental illness which may require treatment.

The investigator, or authorised designee, will allocate then the research participant to a trial treatment arm using one of sixteen (8 per centre) prepared randomisation lists.

The investigator, or authorised designee, will chose the appropriate list based on the participant's centre, HbA1c level (HbA1c < 38mmol/mol or ≥ 38mmol/mol), BMI level (BMI < 30 kg/m2 or ≥ 30kg/m2) and previous response to NB-UVB (achieved remission within 25 exposures during most recent course of NBUVB or not). Those who have not been exposed previously to NBUVB will be placed in the "did not achieve remission within 25 exposures" group.

For research participants allocated randomly to treatment arm A the investigator, or authorised designee, will ask the participant to bring back all used and unused Januvia® tablet packages at each study visit to enable a pill compliance check to be performed.

1st Treatment visit (Visit 3, Week 3 +/- 7 days)

The following assessments will be performed:

1. Completion of quality of life questionnaires by the research participant as detailed in Baseline Visit above;
2. Recording of adverse events;
3. Recording of changes in concomitant medication;
4. Assessment of study drug compliance (pill count);
5. Measurement of weight, blood pressure and heart rate;
6. Assessment of PASI; and
7. Blood sampling for laboratory examination.

2nd Treatment visit (Visit 4, Week 6 +/- 7 days)

The following assessments will be performed:

1. Completion of quality of life questionnaires by the research participant as detailed in Baseline Visit above;
2. Recording of adverse events;
3. Recording of changes in concomitant medication;
4. Assessment of study drug compliance (pill count);
5. Measurement of weight, blood pressure and heart rate;
6. Assessment of PASI; and
7. Blood sampling for laboratory examination.

3rd Treatment visit (Visit 5, Week 12 +/- 7 days)

The following assessments will be performed:

1. Completion of quality of life questionnaires by the research participant as detailed in Baseline Visit above;
2. Recording of adverse events;
3. Recording of changes in concomitant medication;
4. Assessment of study drug compliance (pill count);
5. Measurement of weight, blood pressure and heart rate;
6. Assessment of PASI; and
7. Blood sampling for laboratory examination.

4th Treatment visit (Visit 6, Week 24 +/- 7 days)

The following assessments will be performed:

1. Completion of quality of life questionnaires by the research participant as detailed in Baseline Visit above;
2. Recording of adverse events;
3. Recording of changes in concomitant medication;
4. Assessment of study drug compliance (pill count);
5. Measurement of weight, blood pressure and heart rate;
6. Assessment of PASI; and
7. Blood sampling for laboratory examination. If the participant is willing, and had a skin biopsy performed during visit 2, a skin biopsy will be performed, using sterile technique by an experienced physician, to determine skin immune cell number and skin pro-inflammatory protein level.

1st Follow-Up visit (Visit 7, Week 30 +/- 7 days)

The following assessments will be performed:

1. Completion of quality of life questionnaires by the research participant as detailed in Baseline Visit above;
2. Recording of adverse events;
3. Recording of changes in concomitant medication;
4. Measurement of weight, blood pressure and heart rate;
5. Assessment of PASI; and
6. Blood sampling for laboratory examination.

End of Study visit (Visit 8, Week 36 +/- 7 days)

The following assessments will be performed:

1. Completion of quality of life questionnaires by the research participant as detailed in Baseline Visit above;
2. Recording of adverse events;
3. Recording of changes in concomitant medication;
4. Measurement of weight, blood pressure and heart rate;
5. Performing a urine based pregnancy test (women of child bearing potential only);
6. Assessment of PASI; and
7. Blood sampling for laboratory examination.

Early Withdrawal visit: All research participants who withdraw early from the study will be advised to agree to attend an early withdrawal visit.

There will be a separate section in the CRF to be completed if the research participant withdraws early from the study before week 36.

The following assessments will be performed:

1. Completion of quality of life questionnaires by the research participant as detailed in Baseline Visit above;
2. Recording of adverse events;
3. Recording of changes in concomitant medication;
4. Assessment of study drug compliance (pill count) if appropriate;
5. Measurement of weight, blood pressure and heart rate;
6. Performing a urine based pregnancy test (women of child bearing potential only);
7. Assessment of PASI; and
8. Blood sampling for laboratory parameters.

The research participant's involvement in this study will end following the completion of the End of Study Visit (or Early Withdrawal visit if applicable). Once participants have completed their involvement in this study they will be provided with standard treatment by their usual healthcare providers.

Adverse Events:

Comprehensive assessments of any apparent toxicity experienced by the research participant will be performed throughout the course of the study from the time of participant's signature of informed consent.

Adverse events (AEs) considered related to Study Drug at the End of Study Visit (or Early Withdrawal Visit, if applicable) will be followed until the participant is stable or the AE is resolved or the participant is lost to follow-up.

Any medical condition, or clinically significant laboratory abnormality with an onset date before the Baseline Visit and not related to a protocol-associated procedure, is not an AE. It will be considered to be pre-existing.

Complete and appropriate data on all Adverse Events experienced (observed, volunteered or elicited) during the reporting period will be reported on an ongoing basis in the Adverse Event Form pages of the Case Report Form. The investigator will classify the severity of an adverse event. The investigator will systematically assess the relationship of the adverse event to the investigational medicinal product.

Reporting of Serious Adverse Events (SAEs) Information about all SAEs will be collected and recorded on the SAE Report Form. Each SAE must be reported by the Investigator, or an authorised designee, to the Sponsor within 24 hours of learning of its occurrence.

Medical and scientific judgement will be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalisation, but may jeopardise the research participant or may require intervention to prevent one of the other outcomes listed in the definition above. These will be considered also serious.

Justification of Population and Method of Estimation:

We plan to enrol 120 research participants in total in the two sites. The primary objective of the research project is to determine the change in the psoriasis area and severity index (ΔPASI) during twenty four weeks of treatment with a dipeptidyl peptidase-4 inhibitor (Januvia®, 100mg daily or 50mg daily for participants with moderate kidney disease) in psoriasis patients undergoing narrow-band ultraviolet-B (NB-UVB) light therapy. This will be compared to the ΔPASI of psoriasis patients undergoing NB-UVB light therapy who are allocated randomly to not receive any additional treatment.

Kleinpenning et al have determined previously the effect of two different NB-UVB light therapy regimens on the decrease in PASI three months after completion of a course of NB-UVB light therapy. Three months after cessation of NB-UVB light therapy the decrease in the PASI in those receiving an high-dose regimen was 5.93±4.1compared to baseline. This decrease in PASI was significantly less in the group receiving a low-dose regimen (4.14±2.96, p<0.05).

Based on these data, and assuming a 33% dropout rate, we have calculated that we will require 60 research participants (in each arm) to detect a greater than 33% difference in the ΔPASI with 80% power and a 5% significance level.

Method of Randomisation:

The unit of randomisation will be the individual research participant. After stratification by centre, by HbA1c level (HbA1c < 38mmol/mol or ≥ 38mmol/mol), BMI level (BMI < 30 kg/m2 or ≥ 30 kg/m2) and previous response to NB-UVB (achieved remission within 25 exposures during most recent course of NBUVB or not) 120 research participants will be assigned randomly, in a ratio of 1:1 using blocks of 2, to receive either:

Januvia® tablets; OR No additional treatment.

In order to achieve this we have prepared 8 randomisation lists using a web-based random generator programme. One copy of this document will be used for each centre.

For each participant the investigator, or authorised designee, will chose the appropriate list and will add the participant's identifier to the list in chronological order. This list will be thereby used to determine the study treatment which the participant will receive.

Random allocation will occur at visit 2 (baseline visit) once all screening procedures required at visit 1 (screening visit) have been completed, once it has been confirmed that the participant satisfies all inclusion and exclusion criteria and once the participant completes the three week run-in period.

Identification numbers will be assigned chronologically in consecutive, ascending order.

Independent Ethics Committee (IEC)/Institutional Review Board (IRB) Approval:

Before initiating this study the Study Protocol, Summary of Product Characteristics (SPC), Patient Information Leaflet and Informed Consent Form, applicable advertising, and any other written information to be given to participants will be reviewed and approved by a properly constituted Institutional Review Board/Independent Ethics Committee (IEC/IRB). A signed and dated statement that all documents submitted for review have been approved by the IEC/IRB will be given to the Sponsor or designee before the study can commence at a site. The membership and the constitution of the IEC/IRB who approved the documents will be also supplied to the Sponsor or designee.

Ethical Conduct of the Study:

This study will be carried out in compliance with the Study Protocol and in accordance with the Sponsor/Contract Research Organisations (CROs) Standard Operating Procedures (SOPs). These are designed to ensure adherence to Good Clinical Practice (GCP) guidelines, as described in:

International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Harmonized Tripartite Guidelines for Good Clinical Practice 1996.

European Union (EU) CT Directive 2001/20/EC. GCP Commission Directive 2005/28/EC. Declaration of Helsinki, concerning medical research in humans (1964) including all amendments up to and including the 2008 revision.

National laws. The investigator agrees, when signing the Study Protocol, to adhere to the instructions and procedures described in it and to the principles of GCP to which it conforms.

The regulatory permission to perform the study will be obtained in accordance with applicable regulatory requirements. All ethical and regulatory approvals must be available before a patient is exposed to any study-related procedure, including screening tests to determine eligibility.

Insurance:

In case of any damage or injury occurring to a patient in association with the investigational medicinal product or their participation in the study, the sponsor has insurance which covers the liability of the sponsor, the investigator and other persons involved in the study in compliance with the laws of Ireland.

All investigators are qualified and practicing physicians and are thus insured by the clinical indemnity scheme.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of generalized chronic plaque and/or guttate psoriasis;
2. Are male and female patients aged between 18 and 75 years inclusive;
3. Have a psoriasis area and severity index (PASI) greater than 7 despite use of topical therapies;
4. Are due to undergo NB-UVB light therapy;
5. Have not required systemic psoriasis therapy during the past eight weeks;
6. Are unlikely to require systemic therapy for the duration of clinical trial involvement;
7. Have a negative pregnancy test at screening (women of child bearing potential only); and
8. Are willing to sign voluntarily a statement of informed consent to participate in the study.

Exclusion Criteria:

People with any of the following conditions will be excluded from the study:

1. Photosensitive disorders (lupus erythematosis etc);
2. Diabetes mellitus;
3. Use of medications that can cause photosensitivity;
4. Use of GLP-1 analogue therapy;
5. Conditions that could be made worse by phototherapy (cataract, epilepsy, etc);
6. Allergy or hypersensitivity to Januvia®;
7. Severe kidney disease as defined by a previous diagnosis of chronic kidney disease in the presence of an estimated glomerular filtration rate (eGFR) of less than 30ml/min/1.73m2;
8. Recent (within 8 weeks) receipt of NB-UVB light;
9. Current or recent (within 8 weeks) use of systemic therapy for psoriasis;
10. Severe heart disease as defined by a previous diagnosis of heart disease and a left ventricular ejection fraction which is known to be less than 35% (as measured by echocardiogram or cardiac catheterisation study);
11. Severe lung disease as defined by a previous diagnosis of chronic lung disease and a forced expiratory volume in 1 second (FEV1) or a forced vital capacity (FVC) that is known to be less than 50% that which would be estimated for a person of that age and gender;
12. Severe liver disease as defined by a previous diagnosis of chronic liver disease in the presence of an alanine transferase concentration greater than 150 international units/L (greater than three times the upper limit of the normal reference range);
13. Any other contraindications to Januvia® as stated in its SPC;
14. Female patients of child bearing potential who are pregnant, breastfeeding, or unwilling to practice an acceptable barrier and/or hormonal method of contraception during participation in the study - abstinence will be permitted only if it is in keeping with a person's lifestyle;
15. Any clinically significant chronic disease that might in the opinion of the investigator, interfere with the evaluations or preclude completion of the trial;
16. A current or recent (within the past 4 weeks) acute serious illness, acute psychiatric illness or severe uncontrolled/unstable illness;
17. Previous randomisation into this study;
18. Concurrent participation in another clinical trial; and
19. Participation in another clinical trial during the twelve weeks prior to study entry (i.e. screening visit).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The change in PASI during treatment with sitagliptin for participants with psoriasis undergoing NB-UVB light therapy compared to psoriasis patients undergoing NB-UVB light therapy who are allocated randomly to not receive any additional treatment. | 24 weeks

SECONDARY OUTCOMES:
The incidence of adverse events in the patients treated with sitagliptin and in the patients receiving no additional treatment | 24 and 36 weeks
The change in DLQI in patients receiving treatment with sitagliptin compared to the change in DLQI in patients receiving no additional treatment. | 24 and 36 weeks
  DLQI: dermatology life quality index
The change in PASI over 36 weeks in patients treated with sitagliptin compared to patients receiving no additional treatment. | 36 weeks
The change in blood pressure in patients treated with sitagliptin compared to patients receiving no additional treatment. | 24 and 36 weeks
The change in serum cytokines in patients treated with sitagliptin compared to patients receiving no additional treatment. | 24 and 36 weeks
  Changes in serum concentrations of cytokines (C-reactive protein, interleukin-6 (IL-6), tumour necrosis factor alpha (TNFα) etc) Changes in serum concentrations of hormones (GLP-1, peptide YY (PYY) etc); and Changes in peripheral blood mononuclear cell expression of immune proteins (IL-6, TNFα, IL-10, IL-27 etc).
The incidence of discontinuation of the study investigational medicinal product (IMP). | 24 weeks
The change in HADS in patients receiving treatment with sitagliptin compared to the change in HADS in patients receiving no additional treatment. | 24 and 36 weeks
  HADS: Hospital Anxiety and Depression Scale
The change in HAQ8 in patients receiving treatment with sitagliptin compared to the change in HAQ8 in patients receiving no additional treatment. | 24 and 36 weeks
  HAQ8: Stanford Health Assessment Questionnaire 8-item disability scale
The change in EQ-5D in patients receiving treatment with sitagliptin compared to the change in EQ-5D in patients receiving no additional treatment. | 24 and 36 weeks
  EQ-5D: EuroQOL five item questionnaire
The incidence of achievement of a greater than 50% reduction in PASI from baseline (PASI-50) in patients receiving sitagliptin and in patients receiving no additional treatment. | 36 weeks
The incidence of achievement of a greater than 75% reduction in PASI from baseline (PASI-75) in patients receiving sitagliptin and in patients receiving no additional treatment. | 36 weeks
The incidence of achievement of a greater than 90% reduction in PASI from baseline (PASI-90) in patients receiving sitagliptin and in patients receiving no additional treatment. | 36 weeks
The dosage of narrow-band ultraviolet-B light received by patients receiving sitagliptin and by patients receiving no additional treatment. | 36 weeks
The number of exposures of narrow-band ultraviolet-B light received by patients receiving sitagliptin and by patients receiving no additional treatment. | 36 weeks
The proportion of patients who relapse (PASI greater than 50% of original value) within 36 weeks of commencement of NBUVB light therapy in patients receiving sitagliptin and in patients receiving no additional treatment. | 36 weeks
The times taken to achieve PASI-50, PASI-75, PASI-90 and relapse in patients receiving sitagliptin and in patients receiving no additional treatment. | 36 weeks
The change in glycaemic measures in patients treated with sitagliptin compared to patients receiving no additional treatment. | 24 and 36 weeks
The change in lipid fractions in patients treated with sitagliptin compared to patients receiving no additional treatment. | 24 and 36 weeks
The change in weight in patients treated with sitagliptin compared to patients receiving no additional treatment. | 24 and 36 weeks

OTHER OUTCOMES:
The changes in skin levels of cells in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The genetic, and/or epigenetic, profile that predicts best response to NB-UVB light therapy and to sitagliptin therapy. | Baseline
The changes in expression of cells in skin in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The changes in expression of hormones in skin in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The changes in expression of receptors in skin in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The changes in expression of enzymes in skin in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The changes in expression of immune proteins in skin in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The changes in skin levels of hormones in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The changes in skin levels of receptors in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The changes in skin levels of enzymes in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks
The changes in skin levels of immune proteins in patients treated with sitagliptin and in patients receiving no additional treatment in a sub-group of patients willing to undergo skin biopsies. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kirby, MD FRCPI, Principal Investigator — University College Dublin
Locations (1):
- UCD Clinical Research Centre, St Vincent's University Hospital, Dublin, Ireland

REFERENCES:
- [Result] Schon MP, Boehncke WH. Psoriasis. N Engl J Med. 2005 May 5;352(18):1899-912. doi: 10.1056/NEJMra041320. No abstract available. PMID 15872205
- [Result] Nestle FO, Kaplan DH, Barker J. Psoriasis. N Engl J Med. 2009 Jul 30;361(5):496-509. doi: 10.1056/NEJMra0804595. No abstract available. PMID 19641206
- [Result] Novelli M, Savoia P, Fierro MT, Verrone A, Quaglino P, Bernengo MG. Keratinocytes express dipeptidyl-peptidase IV (CD26) in benign and malignant skin diseases. Br J Dermatol. 1996 Jun;134(6):1052-6. PMID 8763423
- [Result] van Lingen RG, van de Kerkhof PC, Seyger MM, de Jong EM, van Rens DW, Poll MK, Zeeuwen PL, van Erp PE. CD26/dipeptidyl-peptidase IV in psoriatic skin: upregulation and topographical changes. Br J Dermatol. 2008 Jun;158(6):1264-72. doi: 10.1111/j.1365-2133.2008.08515.x. Epub 2008 Mar 29. PMID 18384439
- [Result] Thielitz A, Reinhold D, Vetter R, Bank U, Helmuth M, Hartig R, Wrenger S, Wiswedel I, Lendeckel U, Kahne T, Neubert K, Faust J, Zouboulis CC, Ansorge S, Gollnick H. Inhibitors of dipeptidyl peptidase IV and aminopeptidase N target major pathogenetic steps in acne initiation. J Invest Dermatol. 2007 May;127(5):1042-51. doi: 10.1038/sj.jid.5700439. Epub 2006 Jun 15. PMID 16778789
- [Result] Ohnuma K, Hosono O, Dang NH, Morimoto C. Dipeptidyl peptidase in autoimmune pathophysiology. Adv Clin Chem. 2011;53:51-84. doi: 10.1016/b978-0-12-385855-9.00003-5. PMID 21404914
- [Result] Nishioka T, Shinohara M, Tanimoto N, Kumagai C, Hashimoto K. Sitagliptin, a dipeptidyl peptidase-IV inhibitor, improves psoriasis. Dermatology. 2012;224(1):20-1. doi: 10.1159/000333358. Epub 2011 Nov 1. PMID 22056790
- [Result] Heydendael VM, Spuls PI, Opmeer BC, de Borgie CA, Reitsma JB, Goldschmidt WF, Bossuyt PM, Bos JD, de Rie MA. Methotrexate versus cyclosporine in moderate-to-severe chronic plaque psoriasis. N Engl J Med. 2003 Aug 14;349(7):658-65. doi: 10.1056/NEJMoa021359. PMID 12917302
- [Result] Griffiths CE, Strober BE, van de Kerkhof P, Ho V, Fidelus-Gort R, Yeilding N, Guzzo C, Xia Y, Zhou B, Li S, Dooley LT, Goldstein NH, Menter A; ACCEPT Study Group. Comparison of ustekinumab and etanercept for moderate-to-severe psoriasis. N Engl J Med. 2010 Jan 14;362(2):118-28. doi: 10.1056/NEJMoa0810652. PMID 20071701
- [Result] Pepys MB, Hirschfield GM. C-reactive protein: a critical update. J Clin Invest. 2003 Jun;111(12):1805-12. doi: 10.1172/JCI18921. No abstract available. PMID 12813013
- [Result] Hattori S. Sitagliptin reduces albuminuria in patients with type 2 diabetes. Endocr J. 2011;58(1):69-73. doi: 10.1507/endocrj.k10e-382. Epub 2010 Dec 28. PMID 21206136
- [Result] Derosa G, Maffioli P, Salvadeo SA, Ferrari I, Ragonesi PD, Querci F, Franzetti IG, Gadaleta G, Ciccarelli L, Piccinni MN, D'Angelo A, Cicero AF. Effects of sitagliptin or metformin added to pioglitazone monotherapy in poorly controlled type 2 diabetes mellitus patients. Metabolism. 2010 Jun;59(6):887-95. doi: 10.1016/j.metabol.2009.10.007. Epub 2009 Dec 16. PMID 20015525
- [Result] Williams-Herman D, Engel SS, Round E, Johnson J, Golm GT, Guo H, Musser BJ, Davies MJ, Kaufman KD, Goldstein BJ. Safety and tolerability of sitagliptin in clinical studies: a pooled analysis of data from 10,246 patients with type 2 diabetes. BMC Endocr Disord. 2010 Apr 22;10:7. doi: 10.1186/1472-6823-10-7. PMID 20412573
- [Result] Lamanna C, Monami M, Bartoli N, Zannoni S, Mannucci E. Dipeptidyl peptidase- 4 inhibitors and cardiovascular events: a protective effect? Diabetologia. 2011;54:S109.
- [Result] Chodorowska G, Wojnowska D, Juszkiewicz-Borowiec M. C-reactive protein and alpha2-macroglobulin plasma activity in medium-severe and severe psoriasis. J Eur Acad Dermatol Venereol. 2004 Mar;18(2):180-3. doi: 10.1111/j.1468-3083.2004.00863.x. PMID 15009298
- [Result] Gisondi P, Malerba M, Malara G, Puglisi Guerra A, Sala R, Radaeli A, Calzavara-Pinton P, Girolomoni G. C-reactive protein and markers for thrombophilia in patients with chronic plaque psoriasis. Int J Immunopathol Pharmacol. 2010 Oct-Dec;23(4):1195-202. doi: 10.1177/039463201002300423. PMID 21244768
- [Result] Nisa N, Ahmed Q. High-sensitivity C-reactive protein in psoriasis. Int J Dermatol. 2012 Nov;51(11):1393-4. doi: 10.1111/j.1365-4632.2010.04761.x. Epub 2011 May 30. No abstract available. PMID 21623773
- [Result] Mittal R, Malhotra S, Pandhi P, Kaur I, Dogra S. Efficacy and safety of combination Acitretin and Pioglitazone therapy in patients with moderate to severe chronic plaque-type psoriasis: a randomized, double-blind, placebo-controlled clinical trial. Arch Dermatol. 2009 Apr;145(4):387-93. doi: 10.1001/archdermatol.2009.5. PMID 19380660
- [Result] Drucker DJ, Sherman SI, Gorelick FS, Bergenstal RM, Sherwin RS, Buse JB. Incretin-based therapies for the treatment of type 2 diabetes: evaluation of the risks and benefits. Diabetes Care. 2010 Feb;33(2):428-33. doi: 10.2337/dc09-1499. No abstract available. PMID 20103558
- [Result] Hossler EW, Maroon MS, Mowad CM. Gastric bypass surgery improves psoriasis. J Am Acad Dermatol. 2011 Jul;65(1):198-200. doi: 10.1016/j.jaad.2010.01.001. Epub 2010 Jul 22. PMID 20655127
- [Result] Hogan AE, Tobin AM, Ahern T, Corrigan MA, Gaoatswe G, Jackson R, O'Reilly V, Lynch L, Doherty DG, Moynagh PN, Kirby B, O'Connell J, O'Shea D. Glucagon-like peptide-1 (GLP-1) and the regulation of human invariant natural killer T cells: lessons from obesity, diabetes and psoriasis. Diabetologia. 2011 Nov;54(11):2745-54. doi: 10.1007/s00125-011-2232-3. Epub 2011 Jul 9. PMID 21744074
- [Result] Ahern T, Tobin AM, Corrigan MA, Hogan AE, Kirby B, O'Shea D. Liraglutide Decreases Psoriasis Severity. Irish Journal of Medical Science. 2011;180(Supplement 13):S506.
- [Result] Ahern T, Tobin AM, Corrigan M, Hogan A, Sweeney C, Kirby B, O'Shea D. Glucagon-like peptide-1 analogue therapy for psoriasis patients with obesity and type 2 diabetes: a prospective cohort study. J Eur Acad Dermatol Venereol. 2013 Nov;27(11):1440-3. doi: 10.1111/j.1468-3083.2012.04609.x. Epub 2012 Jun 13. PMID 22691169
- [Result] Monami M, Dicembrini I, Antenore A, Mannucci E. Dipeptidyl peptidase-4 inhibitors and bone fractures: a meta-analysis of randomized clinical trials. Diabetes Care. 2011 Nov;34(11):2474-6. doi: 10.2337/dc11-1099. PMID 22025784
- [Result] Ibbotson SH, Bilsland D, Cox NH, Dawe RS, Diffey B, Edwards C, Farr PM, Ferguson J, Hart G, Hawk J, Lloyd J, Martin C, Moseley H, McKenna K, Rhodes LE, Taylor DK; British Association of Dermatologists. An update and guidance on narrowband ultraviolet B phototherapy: a British Photodermatology Group Workshop Report. Br J Dermatol. 2004 Aug;151(2):283-97. doi: 10.1111/j.1365-2133.2004.06128.x. PMID 15327535
- [Result] Menter A, Korman NJ, Elmets CA, Feldman SR, Gelfand JM, Gordon KB, Gottlieb A, Koo JYM, Lebwohl M, Lim HW, Van Voorhees AS, Beutner KR, Bhushan R. Guidelines of care for the management of psoriasis and psoriatic arthritis: Section 5. Guidelines of care for the treatment of psoriasis with phototherapy and photochemotherapy. J Am Acad Dermatol. 2010 Jan;62(1):114-135. doi: 10.1016/j.jaad.2009.08.026. Epub 2009 Oct 7. PMID 19811850
- [Result] Markham T, Rogers S, Collins P. Narrowband UV-B (TL-01) phototherapy vs oral 8-methoxypsoralen psoralen-UV-A for the treatment of chronic plaque psoriasis. Arch Dermatol. 2003 Mar;139(3):325-8. doi: 10.1001/archderm.139.3.325. PMID 12622624
- [Result] Ryan C, Renfro L, Collins P, Kirby B, Rogers S. Clinical and genetic predictors of response to narrowband ultraviolet B for the treatment of chronic plaque psoriasis. Br J Dermatol. 2010 Nov;163(5):1056-63. doi: 10.1111/j.1365-2133.2010.09985.x. PMID 20716226
- [Result] Kleinpenning MM, Smits T, Boezeman J, van de Kerkhof PC, Evers AW, Gerritsen MJ. Narrowband ultraviolet B therapy in psoriasis: randomized double-blind comparison of high-dose and low-dose irradiation regimens. Br J Dermatol. 2009 Dec;161(6):1351-6. doi: 10.1111/j.1365-2133.2009.09212.x. Epub 2009 Apr 10. PMID 19466961
- [Derived] Lynch M, Ahern TB, Timoney I, Sweeney C, Kelly G, Hughes R, Tobin AM, O'Shea D, Kirby B. Dipeptidyl peptidase-4 inhibition and narrow-band ultraviolet-B light in psoriasis (DINUP): study protocol for a randomised controlled trial. Trials. 2016 Jan 15;17:29. doi: 10.1186/s13063-016-1157-z. PMID 26767505
- See also: A web-based randomization plan generator. — http://www.randomization.com